CLINICAL TRIAL: NCT00452218
Title: Sorafenib Study: Dosing in Patients With Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14636A
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open (Experimental)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 200 mg daily and dose escalated to a maximum of 400 mg twice daily
  Other Names: BAY 43-9006; Nexavar

SUMMARY:
The purpose of this study is to assess the safety and tolerability of sorafenib in patients with PAH already on existing therapy with a prostacyclin [epoprostenol (Flolan)], treprostinil (Remodulin), or iloprost alone, or with or without sildenafil (Viagra/Revatio).

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is an angioproliferative vasculopathy resulting from abnormal endothelial and smooth muscle cell interactions. Idiopathic and familial PAH (formerly known as primary pulmonary hypertension) occurs more often in women than in men, with a median survival of 2.8 years if untreated and a mean age at diagnosis of 35 years. The key features of this vasculopathy causes a progressive narrowing of the pulmonary artery and their branches, resulting in right heart failure and death. Proliferating endothelial cells obliterate medium-sized precapillary arteries, thereby forming the characteristic "plexiform" lesions. When combined with the expansion of both vascular smooth muscle cells and adventitial cells in pulmonary arteries, these observations evoke comparisons to cancer pathobiology. Currently, FDA-approved therapies for PAH such as prostacyclins (epoprostenol, treprostinil, and iloprost), endothelin receptor blockers (bosentan) and phosphodiesterase inhibitors (sildenafil) all produce functional improvement (6 minute walk distance- 6MW) with minimal change in hemodynamic measurements at cardiac catheterization. Only epoprostenol has provided survival benefit with the 5-year survival, remaining at 50% without demonstrable reversal of the vasculopathy. Clearly there is a critical need for novel targets and therapies for PAH.

In this protocol, the principal investigator (PI) will leverage a large PAH referral practice with an established clinical database to assess the potential utility of kinase inhibitors as a new class of agents for protease-activated receptor (PAR). These drugs inhibit processes important to pathological blood vessel branching and growth and have been a focus for the internationally renowned University of Chicago Phase I/II trials unit in oncology led by Dr. Mark Ratain (Co-Investigator). The University of Chicago has had a major role in the drug development of the recently (12/05) FDA-approved drug, sorafenib, for advanced renal carcinoma. Sorafenib inhibits Raf-1 kinase, a regulator of endothelial apoptosis, and inhibits angiogenesis growth factor receptors VEGFR-2, PDGFR-B, and VEGFR-3.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* PAH defined as IPAH, FPAH, or PAH associated with collagen vascular disease
* Baseline 6MW > 150 meters
* PAH as defined by hemodynamics at diagnosis by right heart catheterization defined as: mean PAP > 25 mmHg with a normal PCWP < 15 mm Hg at rest and a PVR > 3 Wood units
* Receiving conventional therapy as clinically indicated (oxygen, diuretics, aldosterone antagonist, calcium channel blockers, digoxin) with dose that is unchanged in the preceding 30 days prior to enrollment. This is excluding anticoagulants (warfarin) as the patient's dose may not be stable if the patient is having a cardiac catheterization at baseline within 30 days of enrollment and warfarin is being held. The dose of warfarin needs to be stable for 7 days or therapeutic with an INR = 2.0
* If on intravenous/subcutaneous prostacyclin at a stable dose > 30 days
* If subjects are on sildenafil, must be at a stable dose > 30 days
* Must have right heart catheterization on prostacyclin + sildenafil within preceding 30 days. Subjects must be on a stable dose of medication within 30 days prior to cardiac catheterization and therefore there can be no dosage changes of the medications between catheterization and baseline
* Must have pulmonary function tests (PFT) within 90 days prior to enrollment: TLC, FEV1, FVC, DLCO
* Women of childbearing years must use adequate contraception (hormonal or barrier method of birth control) prior to enrollment. Subjects need to have a negative serum or urine pregnancy test.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

* PAH associated with all other etiologies: HIV, portopulmonary disease, congenital heart disease
* Subjects with pulmonary hypertension due to thromboembolism, significant interstitial lung disease, chronic obstructive pulmonary disease, congestive heart failure, valvular heart disease
* Subjects with (World Health Organization (WHO) functional Class IV(19)
* Subjects with scleroderma with total lung capacity (TLC) < 60% of predicted within 30 days of screening
* Subjects with significant obstructive lung disease with FEV1/FVC < 80% of predicted
* Subjects with hypotension defined as systolic arterial pressure < 90 mmHg at baseline
* Subjects with hypertension defined as systolic arterial pressure >140 mmHg at baseline or a diastolic arterial pressure > 90 mmHg
* Subjects with impaired renal function defined as creatinine clearance < 30 ml/min as defined by the Cockcroft-Gault formula:

  * Male: creatinine clearance (ml/min) = (140-age) x (body weight in kg)/ (72x serum creatinine in mg/dl);
  * Female: creatinine clearance (ml/min)= 0.85 (140-age) x (body weight in kg)/ (72x serum creatinine in mg/dl)
* Subjects with liver function tests (transaminases (AST/ALT), total bilirubin, and alkaline phosphatase) > 2X normal values
* Subjects with acutely decompensated heart failure or hospitalization within the previous 30 days prior to screening
* Subjects may not be receiving any other investigational agents
* Subjects on endothelin receptor antagonists (bosentan, sitaxsentan, ambrisentan) or chronic arginine supplementation
* Subjects with left ventricular ejection fraction < 45% or left ventricular shortening fraction < 0.2
* Subjects with acute myocardial infarction within 90 days prior to screening
* Subjects with limitations to performance of exercise measures (6MW) due to conditions other than PH associated dyspnea/fatigue
* Subjects taking nitrates for any medical problem
* Subjects taking phosphodiesterase inhibitors (any formulation) for erectile dysfunction
* Subjects with a recent (< 180 days) history of pulmonary embolism verified by ventilation/perfusion scan, angiogram, or spiral CT scan
* Pregnant or lactating women
* Subjects with a history of current drug abuse including alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Monthly 6MW/B | 16 weeks

SECONDARY OUTCOMES:
Efficacy | 16 Weeks
World Health Organization (WHO) function class | 16 weeks
Right heart catheterization | 16 Week
Naughton Balke-Treadmill Test | 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mardi Gomberg, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States